CLINICAL TRIAL: NCT05077644
Title: Mobile Application in the Management of Mild to Moderate Postpartum Depression (PPD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Curio Digital Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CU-T-002
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Post-partum Depression
Keywords: post-partum depression, depression, anxiety, PPD
MeSH Terms: conditions — Depression, Postpartum; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Data from 65 participants (n=50 in this extended study of a piloted user study) will be collected and analyzed to assess the user experience of the Stella (TM) App. Participants will be selected if they have given birth in the four months prior to the study start date, meet eligibility criteria and and have mild-to moderate postpartum depression or have experienced depressive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Participants who use Stella App (Other): Participant experience in using the mobile application and EPDS results
  Interventions: Device: Stella (TM) Mobile Application

INTERVENTIONS:
Device: Stella (TM) Mobile Application — Treatment of mild-to-moderate postpartum depression (PPD) using Cognitive Behavioral Therapy techniques.

SUMMARY:
Primary Objective: Evaluate the user experience with the Stella (TM) app for the management of Postpartum Depression in an observed population for 8 calendar weeks.

DETAILED DESCRIPTION:
Women between 18 and 50 years of age who have had a live birth within 4 months prior to study start date and have a diagnosis of mild to moderate PPD. A total of 65 women residing in the state of New York, New Jersey and Connecticut will be recruited to participate in the study. Patient reported outcomes of mild to moderate depression (using EPDS) will be verified by a behavioral health therapist using the Hamilton Depression Rating Scale (HAM-D).

ELIGIBILITY:
Inclusion Criteria:

1. Participants residing in the states of New York, New Jersey or Connecticut and must be able to read, write, and speak English, and provide written informed consent prior to enrollment
2. Participants must be between 18 and 50 years of age
3. Participants must have given live birth within the 4 months prior to the start of study
4. Participants diagnosed with mild to moderate postpartum depression (as assessed by a clinician upon enrollment) and have scored between 9 and 21 on the Edinburgh Postnatal Depression Scale (EPDS) during screening
5. Participants must answer "0/Never" or "1/Hardly Ever" to the self-harm question on EPDS (Question #10)
6. Participants must be willing to use a mobile app and own an iOS enabled mobile phone
7. Participants must have wireless internet connectivity in the home and be willing to connect devices to their home Wi-Fi network.

Exclusion Criteria:

1. Participants who do not reside in the states of New York, New Jersey or Connecticut
2. Participants who are not able to read, write, and speak English, and provide written informed consent prior to enrollment
3. Participants less than 18 and more than 50 years of age
4. Participants who have not given birth within the 4 months prior to the start of study OR did not have a live birth in the last 4 months
5. Participants who have not been diagnosed with postpartum depression upon clinical assessment OR do not have a score of between 9 and 21 on the EPDS
6. Participants with a positive (2 or 3) answer on the EPDS self-harm question (Question #10)
7. Participants with Serious Mental Illnesses (SMIs), severe depression, or cognitive impairments

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult females who delivered live births in the 4 months prior to study start and reported depressive symptoms after child birth
Enrollment: 65 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in level of depression as measured by Edinburgh Postpartum Depression (EPDS) | 8 week period
  Evaluation of difference in mean change in EDPS at week 8 from baseline assessment. EPDS evaluated every 2 weeks from baseline to week 8

SECONDARY OUTCOMES:
Proportion of women who reported App use for daily mood, sleep and activities of daily living | 8 week period
  Summary reported of daily mood, hours of sleep and activities of daily living as identified through the mobile application

CONTACTS AND LOCATIONS:
Overall Officials: Stan Kachnowski, MPA, PhD, Principal Investigator — Healthcare Innovation Technology Lab; Sarah Chokshi, DrPH, Study Director — Healthcare Innovation Technology Lab
Locations (1):
- HITLAB, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No